CLINICAL TRIAL: NCT03333876
Title: In Home Assessment of Three Anti-Snoring Devices, a Cross Over Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Respironics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SRC-AI-SilentNight-10090
Record Dates: First submitted 2017-10-30; First posted 2017-11-07 (Actual); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Snoring
MeSH Terms: conditions — Snoring | interventions — Mandibular Advancement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Nasal Dilator (Active Comparator): Nasal dilators have been used to treat snoring and sleep apnea. Many studies focus on external nasal dilators like Breathe Right Strips. These interventions largely were not effective in treating OSA. However, there is some evidence to suggest internal to the nose dilators (like Mute) may work to reduce snoring
  Interventions: Device: Nasal Dilator
- Mandibular Advancement (Active Comparator): Mandibular advancement devices have shown to be effective, but not necessarily acceptable to primary snorers.
  Interventions: Device: Mandibular Advancement
- Positional Therapy (Active Comparator): Studies have shown mixed results for positional therapy as a whole. Braver and Block reported that foam wedges used to keep patients in a lateral position were not effective in reducing snoring in 20 individuals.
  Interventions: Device: Positional Therapy

INTERVENTIONS:
Device: Nasal Dilator — Mute is a pair of nasal dilators that fit snugly in the nose of the snorer dilating the nostrils to help reduce or eliminate snoring. This is an over-the-counter (OTC) product and is cleared by FDA for use in the United States. The introduction video for Mute is located at http://mutesnoring.com/how-to-use/.
  Arms: Nasal Dilator
Device: Mandibular Advancement — For purposes of this trial, we will be using an investigational myTAP V, which is not available for commercial use. The changes from the released product are: a vertical offset (+3mm) has been added to the design of the adjustment post and mechanism to improve overall comfort.
  myTAPTM is a mandibular advancement device used for snoring relief. The product requires a prescription and is cleared by FDA for use in the United States.
  Arms: Mandibular Advancement
Device: Positional Therapy — Sleep Positional Trainer (SPT) is a small device worn around the chest with an ergonomic band that continuously monitors the sleep position of the snorer. When the snorer is supine, it emits a gentle vibration to remind them to turn to the side to help reduce or eliminate their snoring.
  Arms: Positional Therapy

SUMMARY:
Silent Night is a solution for primary snorers to guide them to the proper anti-snoring solution. It consists of a mobile application, which had an intake questionnaire, guides users to one of three anti-snoring solutions; a nasal dilator called, Mute (Rhinomed, Australia), a mandibular advancement device called myTAP V (Airway Management, Austin, TX) and a Sleep Positional Trainer SPT (SPT) (NightBalance, Netherlands). The Silent Night app also records snoring through the night and provides feedback to the user via a "snore score."

DETAILED DESCRIPTION:
Silent Night is a solution for primary snorers to guide them to the proper anti-snoring solution. It consists of a mobile application, which had an intake questionnaire, guides users to one of three anti-snoring solutions; a nasal dilator called, Mute (Rhinomed, Australia), a mandibular advancement device called myTAP V (Airway Management, Austin, TX) and a Sleep Positional Trainer SPT (SPT) (NightBalance, Netherlands). The Silent Night app also records snoring through the night and provides feedback to the user via a "snore score."

The objective of this trial is twofold. First, each of the interventions to be studied are known to be effective for snoring cessation. However, each is not fully effective in the total population. Their effectiveness is predicated on how an individual snores and where the snore anatomically originates. I.e. if someone position ally snores because their tongue moves back in their mouth, it is unlikely a nasal dilator will work for that individual. In order to improve the SilentNight recommendation algorithm more information needs to be gathered. By asking a battery of questions of a snorer, and having them trial all three snoring solutions it may be possible to understand the comparative effectiveness of each solution, the user acceptance of each solution and which questions should be used to discern what solution will work best for a given individual.

The second objective is to collect "in the wild" audio of snoring. The goal of this data collection, is to identify unique characteristics in the sound recording. These paired with the answers to the intake questions, and the relative effectiveness of the three anti-snoring solutions could phenotype the snore and snorer. This audio data could also be used to develop or refine a "snore score", a semi-objective assessment of snoring audio.

To accomplish these goals, a feasibility, crossover, in home study will be conducted. Up to 30 couples will be recruited to try each of the anti-snoring solutions over an approximately 5 week period. The participant couples will consist of a snorer and a bed partner. The snorer will use the three solutions (1 week for Mute, 2 weeks for myTAP and SPT) and give feedback on the devices, and sleep quality. The bed partner will also provide feedback on their sleep quality, the loudness of snoring and their perception of the device (as a non-user). They will also record bedroom sound during each night of the trial, including a baseline period where no snoring will take place. Each morning the bed partner will rate the snoring severity.

The primary endpoint will be the daily rating of snoring severity as rated by the bed partner. The daily responses will be averaged on a weekly basis. Due to titration and acclimation during the first 9 nights of use nights 10-14 of myTAP V and SPT use will be compared to the week of Mute use. If formal statistical comparisons are performed, continuous data will be compared between the three therapies using repeated-measures ANOVA or the non-parametric Friedman Test, depending on the distributions of the endpoints. If an overall significant effect is observed, post-hoc pairwise tests will be done with a suitable adjustment for multiple comparisons. Categorical data will be compared between therapies using the Cochran's Q test.

ELIGIBILITY:
Inclusion Criteria (Snorer):

* Adults aged 21 to 55
* Able and willing to provide written informed consent
* Able to read and understand English
* History of snoring for more than 6 months (by self-report).
* Sleep with a bed partner for at least 4 nights per week (by self-report).
* Told by bed partner that snoring frequently disturbs his or her sleep (by self-report).
* Have seen a dentist within 12 months (by self-report).
* Willing to not use any anti-snoring aids that are not associated with the study (by self-report).
* Has purchased or used or bed partner has purchased an anti-snoring product in the past (by self-report) [These individuals may be included in the study if recruitment timeline dictates it]

Exclusion Criteria (Snorer):

* Scored higher than a 9 on the Modified Snore Scale Score (MSSS>9)
* Scored higher than a 6 on the OSA 50 screener (OSA50>6)
* The presence of physical or mental limitations that would limit the ability to use the anti-snoring solutions.
* Any unstable medical condition like congestive heart failure, neuromuscular disease, renal failure, or cancer (as determined by self-report and reviewed by the study PI).
* Any severe respiratory condition (like an exacerbation of Chronic Obstructive Pulmonary Disease, bronchitis, sinusitis, respiratory failure or insufficiency or patients requiring oxygen therapy).
* Known history of Obstructive Sleep Apnea (OSA) or Central Sleep Apnea Syndrome (by self-report)
* Only able to sleep in the supine (flat on one's back) position (by self-report).
* Actively suffering from an upper respiratory infection (by self-report).
* Have a planned medical or dental procedure involving the head, neck, face (eyes, ears, nose, teeth, mouth), or lungs during the trial period (by self-report).
* Under active treatment for an active dental problem by a dentist or orthodontist
* Have one or more of the following dental issues (by self-report)

  * Removable dentures or bridges.
  * Temporary crowns, loose teeth, loose crowns, loose fillings, or broken teeth
  * Less than 8 natural, healthy teeth in each dental arch (upper and lower teeth)
  * Dental braces
  * TemporoMandibular Joint (TMJ) issues

Inclusion Criteria (Bed Partner):

* Adults aged 21 to 70
* Able and willing to provide written informed consent
* Able to read and understand English
* Rates sleep disturbance caused by partner's snoring greater than or equal to 4 on a scale of 1-10
* Rates level of snoring volume greater than or equal to 7 on a scale of 1-10
* Willing to sleep in same room as snorer during the study period (by self -report).
* Willing to not start any new over-the-counter or prescription sleep medication including sedatives and hypnotics during the study period (by self-report).

Exclusion Criteria (Bed Partner):

• Told by bed partner that their snoring frequently disturbs his or her sleep (by self-report).

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2017-12-03 (Actual); Study Completion 2017-12-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Philips Respironics, Murrysville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Coded data will be shared with the Philips Research in the Netherlands.
Supporting Information: Study Protocol, ICF
Time Frame: At close of the data collection period that data will be available for analysis. The coded data will be available indefinitely
Access Criteria: Those that have access will be trained to Philips procedures.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 58 participants at one site were consented in October 2017 in Pittsburgh, Pennsylvania. 29 were snorers, 29 were bed partners.
Pre-assignment Details: Of the 29 couples, 2 participants screened out. Therefore 27 participants started the study.
Units Other Than Participants: partners
Groups:
- All Study Participants: All study participants that consented are included in the participant flow.
Period: Screening Period
Arm/Group | All Study Participants
Started | 58; 29 partners
Completed | 54; 27 partners
Not Completed | 4; 2 partners
Not completed — Screen Failure | 4
Period: Nasal Dilator
Arm/Group | All Study Participants
Started | 54; 27 partners
Completed | 48; 24 partners
Not Completed | 6; 3 partners
Not completed — Bed Partner Lost to follow up | 6
Period: Mandibular Advancement
Arm/Group | All Study Participants
Started | 54; 27 partners
Completed | 50; 25 partners
Not Completed | 4; 2 partners
Not completed — Adverse Event | 2
Not completed — Product Damage | 2
Period: Positional Therapy
Arm/Group | All Study Participants
Started | 54; 27 partners
Completed | 54; 27 partners
Not Completed | 0; 0 partners

BASELINE CHARACTERISTICS:
Population: This is all participants that were consented and eligible to participant in the study, all baseline demographics include snorer and bed partner with the exception of neck circumference and Body Mass Index (BMI).
Groups:
- Snorers: All participants that entered the study that were considered snorers.
- Bed Partners: All participants that entered the study that were considered bed partners.
- Total: Total of all reporting groups
Arm/Group | Snorers | Bed Partners | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 29 | 58
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (7.5) | 43.8 (8.3) | 43.7 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 16 | 25
  Male | 20 | 13 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 28 | 28 | 56
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 23 | 24 | 47
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 29 | 29 | 58
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: This only includes snorers. As BMI is an important data element for the snoring group. However, provides no value for bed partner.
  This also excludes the two participants there were found not eligible for the study.
  kg/m^2
    number analyzed (Participants) | 27 | 0 | 27
    (all) | 31.1 (6.5) |  | 31.1 (6.5)
Neck Circumference [Mean (Standard Deviation); unit: inches] — Population: This only includes snorers. As Neck Circumference is an important data element for the snoring group. However, provides no value for bed partner.
  This also excludes the two participants there were found not eligible for the study.
  inches
    number analyzed (Participants) | 29 | 0 | 29
    (all) | 16 (1.5) |  | 16 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Bed Partners' Rating of Sleep Disturbance Due to Partner Snoring
Description: Bed partner subjective feedback based upon a 0 to 10 scale of "how much did your partner's snoring disturb your sleep last night." 0 was the worst, 10 was the best. This is was evaluated at the end of each period.
Time Frame: 5 weeks
Population: This includes all bed partners that completed the subjective feedback survey.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Nasal Dilator: Nasal dilators have been used to treat snoring and sleep apnea. Many studies focus on external nasal dilators like Breathe Right Strips. These interventions largely were not effective in treating Obstructive Sleep Apnea (OSA). However, there is some evidence to suggest internal to the nose dilators (like Mute) may work to reduce snoring.
  Nasal Dilator: Mute is a pair of nasal dilators that fit snugly in the nose of the snorer dilating the nostrils to help reduce or eliminate snoring. This is an over-the-counter (OTC) product and is cleared by FDA for use in the United States. The introduction video for Mute is located at http://mutesnoring.com/how-to-use/.
- Mandibular Advancement: Mandibular advancement devices have shown to be effective, but not necessarily acceptable to primary snorers.
  Mandibular Advancement: For purposes of this trial, we will be using an investigational myTAP V, which is not available for commercial use. The changes from the released product are: a vertical offset (+3mm) has been added to the design of the adjustment post and mechanism to improve overall comfort.
  myTAPTM is a mandibular advancement device used for snoring relief. The product requires a prescription and is cleared by FDA for use in the United States.
- Positional Therapy: Positional Therapy was conducted with a Sleep Positional Trainer (SPT) is a small device worn around the chest with an ergonomic band that continuously monitors the sleep position of the snorer. When the snorer is supine, it emits a gentle vibration to remind them to turn to the side to help reduce or eliminate their snoring.
Arm/Group | Nasal Dilator | Mandibular Advancement | Positional Therapy
Number analyzed (Participants) | 24 | 25 | 27
units on a scale | 5.0 (1.6) | 3.8 (2.2) | 4.4 (2.5)
Statistical Analysis 1: Comparison: Nasal Dilator vs Mandibular Advancement vs Positional Therapy; Each group was compared to baseline; Test type: Superiority; p < .001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Users Acceptance of Each Solution
Description: A star rating based on a 1 -5 scale, overall customer satisfaction with the product (0 to 10 scale), likeliness to buy the product (0 to 10 scale), likeliness to recommend purchase (0 to 10 scale). For the Star rating 1 is the worst, 5 is the best. For the 0 to 10 scale, 0 is the worst, 10 is the best. This was the average acceptance of all users.
Time Frame: 5 weeks
Population: All snorers were included in the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nasal Dilator | Mandibular Advancement | Positional Therapy
Number analyzed (Participants) | 27 | 27 | 27
units on a scale
  Star Rating | 3.4 (0.9) | 2.7 (1.2) | 3.1 (1.1)
  overall customer satisfaction with the product | 6.3 (1.8) | 4.4 (3.3) | 5.5 (2.4)
  likeliness to buy the product | 6.4 (2.7) | 4.1 (3.6) | 5.3 (3.1)

3. Secondary Outcome: Understand User Acceptance of the Bed Partner of Each Solution
Description: likeliness to recommend purchase (0 to 10 scale). 0 is the worst, 10 is the best.
Time Frame: 5 weeks
Population: All bed partners that completed the final survey were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nasal Dilator | Mandibular Advancement | Positional Therapy
Number analyzed (Participants) | 25 | 26 | 27
units on a scale | 4.4 (3.2) | 4.6 (4.0) | 5.4 (3.4)

4. Secondary Outcome: Overall Satisfaction of the Bed Partner of Each Solution
Description: Overall Satisfaction of the Solution from the bed partner (0 to 10 scale). 0 is the worst, 10 is the best.
Time Frame: 5 weeks
Population: All bed partners that completed the final survey were included in the analysis. Not all bed partners completed the final survey.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nasal Dilator | Mandibular Advancement | Positional Therapy
Number analyzed (Participants) | 24 | 26 | 27
units on a scale | 5.0 (3.3) | 5.3 (3.6) | 6.6 (2.7)

5. Secondary Outcome: Total Number of Audio Recordings
Description: Total number of Audio recordings of snoring in different individuals in a baseline setting and using various anti-snoring solutions.
Time Frame: Baseline and 5 weeks
Population: All participants that entered the study had recordings. This record just includes snorer records, not bed partner.
  12 recording could not be counted as they were not classified correctly by participants. Additional baseline nights were recorded by participants because of baseline extension or recordings in between device use.
Measure: Number; unit: audio recordings
Groups:
- Baseline: All participants that entered the study were to complete a baseline period of 3 nights in which no intervention was used, but sleep was recorded.
Arm/Group | Baseline | Nasal Dilator | Mandibular Advancement | Positional Therapy
Number analyzed (Participants) | 27 | 24 | 26 | 27
audio recordings | 113 | 168 | 328 | 308

ADVERSE EVENTS:
Time Frame: All adverse events were collected over a 5 week period on the snorer as the snorer was trying different devices.
Arm/Group | Nasal Dilator | Mandibular Advancement | Positional Therapy
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 0/27 | 3/27 | 0/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nasal Dilator (N=27) | Mandibular Advancement (N=27) | Positional Therapy (N=27)
Jaw Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0) — 3 participants complained of Jaw Pain/Discomfort/Popping

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-14): https://cdn.clinicaltrials.gov/large-docs/76/NCT03333876/Prot_SAP_000.pdf